CLINICAL TRIAL: NCT02553057
Title: Low Tidal Volume for Lung Protection During Anesthesia of Laparoscopic Surgery in Trendlenburg Position
Acronym: lapVent
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: AlRefaey Kandeel (Other)
Responsible Party: Sponsor-Investigator, AlRefaey Kandeel, Dr, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DrSamah
Record Dates: First submitted 2015-09-15; First posted 2015-09-17 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Intraoperative Mechanical Ventilation
MeSH Terms: interventions — Respiration, Artificial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Active Comparator): mechanical ventilation with Tidal volume 4 ml/kg and PEEP 8-10 cm H2o
  Interventions: Device: mechanical ventilation
- Group2 (Active Comparator): mechanical ventilation with Tidal volume 6 ml/kg and PEEP 8-10 cm H2o
  Interventions: Device: mechanical ventilation
- Group 3 (Active Comparator): mechanical ventilation with Tidal volume 8 ml/kg and PEEP 8-10 cm H2o
  Interventions: Device: mechanical ventilation

INTERVENTIONS:
Device: mechanical ventilation

SUMMARY:
Mechanical ventilation of patients undergoing laparoscopic surgery may induce lung injury. Since lung protective ventilation has been recommended during anesthesia to prevent ongoing lung injury, so in our study the investigators will compare three different lung protective strategies regarding their lung protective effect measured by the incidence of postoperative pulmonary complications, perioperative oxygenation and postoperative inflammatory mediator release.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing laparoscopic colorectal or gynaecologic surgery with expected time more than two hours

Exclusion Criteria:

* refusal, preoperative pulmonary disease

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
postoperative pulmonary complications | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university, Al Mansurah, Dkahleya, Egypt